CLINICAL TRIAL: NCT05754515
Title: Evaluation of Oxygenation Parameters in Patients Undergoing Rhinoplasty Under General Anesthesia
Status: Completed | Type: Observational
Sponsor: Duzce University (Other)
Responsible Party: Sponsor
Other Study IDs: PaO2 /FiO2 ratio for TCI
Record Dates: First submitted 2022-10-24; First posted 2023-03-03 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Anesthesia; Functional
Keywords: target controlled anesthesia; oxygenation; inhalation anesthesia
MeSH Terms: interventions — Transcobalamins; Population Groups; Anesthesia, Inhalation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- target controlled infusion (TCI) group: Propofol and remifentanil will be used in TCI anesthesia, and while the patient is under adequate sedation (BIS40-60), muscle relaxation will be provided with 0.6 mg/kg rocurium bromide. While applying TCI anesthesia, the device will use the Minto model for Remifentanil infusion and the Schnider model for Propofol infusion.
  Interventions: Procedure: target controlled infusion (TCI) group
- inhalation anesthesia (IA) groups: During anesthesia induction of patients receiving inhalation anesthesia, 60 mg 2% lidocaine, 2 mg/kg propofol, 0.6 mg/kg rocuronium bromide and 1 mcg/kg fentanyl will be used. Desflurane will be used with a minimum alveolar concentration of 1 and for additional intraoperative sedation. remifentanil will be given between 0.05 and 0.2mcg/kg/min according to the patient's needs.

INTERVENTIONS:
Procedure: target controlled infusion (TCI) group — Patients in the TCI group will be anesthetized with propofol and remifentanil throughout the operation.
  Patients included in the inhalation anesthesia group will be anesthetized with desflurane and remifentanil with a bispectral index of 40-60 throughout the operation.
  Other Names: inhalation anesthesia (IA) group
  Groups: target controlled infusion (TCI) group

SUMMARY:
The investigators are planning to compare the oxygenation values (Pao2/fio2, lactate etc.) in patients who underwent TCI and inhalation anesthesia in rhinoplasty operation.

DETAILED DESCRIPTION:
Total intravenous anesthesia (TIVA) is a common anesthesia method used today as an alternative to inhalation anesthesia. Loss of consciousness is two important components of general anesthesia, in order to give the patient safe analgesia and not to remember any adverse events related to the operation. While the depth of anesthesia can be controlled by monitoring the minimum alveolar concentration (MAK) in the ventilator devices in the operating room we use modernly, there was no more objective method than measuring the plasma level of drugs in intravenous anesthesia. The schemes created by the anesthetists according to plasma drug levels were used when administering total intravenous anesthesia. Target Controlled Anesthesia (TCI) devices, on the other hand, are pumps that have been used more frequently recently and that can deliver the required blood concentration of a drug in bolus and infusion form according to pharmacokinetics models calculated with personal data. In TCI anesthesia, intravenous infusion of anesthetics provides a more stable drug concentration in the plasma and at the site of action compared to repeated bolus techniques. Thus, it is ensured that the drug remains in the therapeutic range, avoiding the consequences such as over- or under-administration of the drugs. The subject of the study is to determine which of the 2 routinely used methods in rhinoplasty operations affects respiratory functions less.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years and younger than 60 years of age who will be operated under general anesthesia
* Patients in I, II risk groups according to the American Society of Anesthesiologists (ASA) classification

Exclusion Criteria:

* ASA III and above patients
* Patients for whom Intensive Care Unit (ICU) indication is prescribed
* Chronic obstructive pulmonary disease
* Having a personal or family history of malignant hyperthermia,
* morbid obesity
* Alcohol or drug addiction
* Have a history of liver or kidney disease
* Coronary artery disease or heart failure
* Anemia
* Hemoglobinopathy
* Sepsis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients over the age of 18 who will undergo general anesthesia will be included in the study.
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
oxygen concentration change throughout the operation | 6 periods; 0. basal blood gas(preoperation), 5 min after intubation, 2 hours after intubation, 5 minutes before extubation, 8 hours after extubation
  In both general anesthesia methods, blood gas measurements will be made at certain intervals, and pao2 /fio2 in percent (%) ratio will be recorded.
tissue oxygen use as lactate change throughout the operation | 6 periods; 0. basal blood gas(preoperation), 5 min after intubation, 2 hours after intubation, 5 minutes before extubation, 8hours after extubation
  In both general anesthesia methods, blood gas measurements will be made at certain intervals serum lactat values mg/dl ratio will be recorded.
airway pressures throughout the operation | during the operation
  Airway pressures in cmH2O will be recorded during both anesthesia methods applied throughout the operation.
lung compliance throughout the operation | during the operation
  The lung compliance in in ml/cmH2O will be recorded during both anesthesia methods applied throughout the operation.

SECONDARY OUTCOMES:
Nausea | Postoperative 24 hour
  Postoperative nausea, vomiting, recovery time from anesthesia will be recorded.
vomiting | Postoperative 24. hour
  Postoperative vomiting, recovery time from anesthesia will be recorded.
recovery time | Postoperative 24 hour
  Postoperative recovery time from anesthesia will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: yavuz demiraran, Study Director — Duzce Univercity Anesthesiogly department
Locations (1):
- Gizem Demir Şenoğlu, Düzce, Düzce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
In accordance with the personal data protection law numbered 6698 dated 24.03.2016 in the constitution of the Republic of Turkey, personal information must be stored and protected only by the people conducting the study.